CLINICAL TRIAL: NCT02731885
Title: An Open, Randomized Study, to Investigate the Potential Food Effect on Pharmacokinetic Parameters of ABX464 Administered Orally to Healthy Male Subjects
Brief Title: Food Effect on Pharmacokinetic Parameters of ABX464
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abivax S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ABX464-FE-001
Record Dates: First submitted 2016-03-25; First posted 2016-04-08 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — ABX464

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasted Conditions (Experimental): 50mg of ABX464 (two 25mg capsules) /Fasted
  Interventions: Drug: ABX464 Single dose; Drug: ABX464 Repeated dose
- Fed Conditions (Experimental): 50mg of ABX464 (two 25mg capsules) /Fed
  Interventions: Drug: ABX464 Single dose; Drug: ABX464 Repeated dose

INTERVENTIONS:
Drug: ABX464 Single dose — Two-periods, subjects received a single dose of 50mg of ABX464 in fed and fasted condition, separated by a wash-out period of at least 45 days.
Drug: ABX464 Repeated dose — Subjects received 50mg of ABX464 every 3 days during 10 days in fasted or fed condition.

SUMMARY:
The goal of this study is to determine the impact of the food on the absorption of the ABX464.

DETAILED DESCRIPTION:
This is a phase I, single-center, open-label, two-treatment, food-effect, randomized study in 40 healthy Caucasian male subjects in order to determine the impact of the food on the absorption of the ABX464.

The two different treatments are the followings:

* Treatment A = 50mg of ABX464 (two 25mg capsules) /Fasted
* Treatment B = 50mg of ABX464 (two 25mg capsules) / Fed

This study consists of two groups:

* Group 1 - single dose assessments, two-period, two-treatment, cross-over: 20 subjects will receive a single dose of 50mg of ABX464 in fed and fasted condition, separated by a wash-out period of at least 45 days.
* Group 2 - multiple dose assessments: 20 subjects will receive 50mg of ABX464 every 3 days during 10 days in fasted or fed condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian male subjects, 18-55 years of age
* Body Mass Index (BMI) of 17-28 kg/m².
* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination)
* Normal vital signs after 10 minutes resting in supine position:

  90 mmHg < systolic blood pressure < 140 mmHg, 50 mmHg < diastolic blood pressure < 90 mmHg, 40 bpm < heart rate < 100 bpm.
* Normal automatic 12-lead ECG (incomplete right bundle branch block can be accepted) or judged as non clinically significant.
* Clinical laboratory tests (hematology, blood chemistry, and urinalysis) must be within normal limits or clinically acceptable to Investigator and Sponsor.
* Subjects must be willing to give written informed consent prior to study enrollment and be able to adhere to restrictions and examination schedules.

Exclusion Criteria:

* Individuals with a history of any significant medical disorder which requires a physician's care (cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic, hematological, neurologic, psychiatric, systemic, or infectious disease; any acute infectious disease or signs of acute illness)
* Frequent headaches and / or migraine, recurrent nausea and / or vomiting (more than twice a month).
* Presence or history of drug allergy, or allergic disease diagnosed and treated by a physician.
* Individuals who have a history of any clinically significant local or systemic infectious disease within 4 weeks prior to drug administration.
* Any individual who does not comply with the requirement that he should not have used any drugs other than paracetamol for at least 2 weeks prior to the study nor alcohol within 48 hours prior to drug administration.
* Individuals who are positive for hepatitis B virus, hepatitis C virus or HIV.
* History or presence of drug or alcohol abuse (positive urine drug screen, positive alcohol breath test).
* Smoking more than 5 cigarettes or equivalent / day, unable to stop smoking during the study.
* Excessive consumption of beverages with xanthine bases (> 4 cups or glasses / day).
* Subject who will likely be unable to eat entirely the standard high fat breakfast within the allocated time.
* Individuals who have donated blood within the preceding 3 months.
* Individuals who refuse to use an effective method of contraception from the beginning of the study and until 3 months after dosing.
* Individuals with forfeiture of freedom by an administrative or legal obligation or under guardianship

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of single oral dose of 50mg of ABX464 in fed or fasted condition. | 45 days
Peak Plasma Concentration (Cmax) of single oral dose of 50mg of ABX464 in fed or fasted condition. | 45 days

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of repeated doses of 50 mg of ABX464 in fed or fasted conditions | 10 days
Peak Plasma Concentration (Cmax) of repeated doses of 50 mg of ABX464 in fed or fasted conditions | 10 days
Number of Subjects with treatment-related adverse events as assessed by CTCAE v4.0 | Up to 45 days

CONTACTS AND LOCATIONS:
Locations (1):
- CAP Research, Sayed Hossen Road, Phoenix, Mauritius

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Scherrer D, Rouzier R, Cardona M, Barrett PN, Steens JM, Gineste P, Murphy RL, Tazi J, Ehrlich HJ. Randomized Trial of Food Effect on Pharmacokinetic Parameters of ABX464 Administered Orally to Healthy Male Subjects. Antimicrob Agents Chemother. 2016 Dec 27;61(1):e01288-16. doi: 10.1128/AAC.01288-16. Print 2017 Jan. PMID 27799203